CLINICAL TRIAL: NCT02324686
Title: Vitamin K Supplementation to Improve INR Stability in Patients on Hemodialysis Taking Warfarin for Atrial Fibrillation
Brief Title: Vitamin K Supplementation in Patients on Hemodialysis
Acronym: VISTA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-8200
Record Dates: First submitted 2014-12-19; First posted 2014-12-24 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2016-05

CONDITIONS: End Stage Renal Failure on Dialysis; Atrial Fibrillation
Keywords: Warfarin; International Normalized Ratio; Vitamin K
MeSH Terms: conditions — Atrial Fibrillation | interventions — Vitamin K 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vitamin K1 (Other): Vitamin K1 400 mcg orally three times a week on dialysis days for four months
  Interventions: Drug: vitamin K1

INTERVENTIONS:
Drug: vitamin K1 — Vitamin K1 400 mcg orally three times a week on dialysis days for four months
  Other Names: phytonadione

SUMMARY:
The purpose of this study is to determine whether vitamin K supplementation will improve anticoagulation control in patients on hemodialysis taking warfarin for atrial fibrillation. Patients who participate will receive vitamin K1 three times a week on dialysis days for a period of four months. INR levels collected during this period will be compared to the four month period prior to receiving the vitamin K1 to determine if vitamin K improves the standard deviation of INRs and time in therapeutic range.

DETAILED DESCRIPTION:
Patients on hemodialysis with atrial fibrillation are at increased risk of stroke. These patients often take warfarin to reduce this risk. Warfarin is a drug that is used to prevent clots in the bloodstream. The dose of warfarin varies from person to person, and its effect is measured using a blood test called the international normalized ratio (INR). In most patients with atrial fibrillation the goal is to keep the INR between 2 and 3. Patients on hemodialysis often have unstable INR levels. Vitamin K supplementation has been shown to improve INR control in patients on warfarin but has not yet been studied in hemodialysis patients.

In this study, patients on hemodialysis receiving warfarin for atrial fibrillation will receive vitamin K 400 mcg orally three times a week on dialysis days for 4 months. INR levels in the four months before and the four months while receiving vitamin K will be reviewed.

The primary end point will look at INR stability and be measured by calculating the standard deviation of INR values before and after receiving vitamin K. The goal of this study is to determine whether vitamin K supplementation improves INR control in patients on hemodialysis taking warfarin for atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* greater than 18 years of age
* Receiving in-house hemodialysis for at least 6 months
* Previously diagnosed with atrial fibrillation
* On warfarin for at least 6 months with a target INR of 2-3

Exclusion Criteria:

* are unable to provide informed consent
* have a mechanical heart valve
* are receiving supplements containing vitamin K
* have a known hypersensitivity to vitamin K

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-01; Primary Completion 2017-12-18 (Actual); Study Completion 2017-12-18 (Actual)

PRIMARY OUTCOMES:
INR stability (standard deviation of INR values) | 4 months before and 4 months after intervention
  standard deviation of INR values, 4 months before and 4 months after the intervention

SECONDARY OUTCOMES:
Time in Therapeutic Range (Percentage of time INR levels within range) | 4 months before and 4 months after intervention
  , 4 months before and 4 months after the intervention
Adverse events | 4 months before and 4 months after intervention
  Number and types of thromboembolic and bleeding complications, 4 months before and 4 months after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Marisa Battistella, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
When the study is complete aggregate data of the study will be published and shared. Individual participant data that may identify participants will not be shared. If a participant requests information on his/her individual participant data, it will be provided to the requesting participant.

REFERENCES:
- [Background] Reinecke H, Engelbertz C, Schabitz WR. Preventing stroke in patients with chronic kidney disease and atrial fibrillation: benefit and risks of old and new oral anticoagulants. Stroke. 2013 Oct;44(10):2935-41. doi: 10.1161/STROKEAHA.113.001701. Epub 2013 Sep 5. No abstract available. PMID 24008579
- [Background] Sood MM, Komenda P, Sood AR, Rigatto C, Bueti J. The intersection of risk and benefit: is warfarin anticoagulation suitable for atrial fibrillation in patients on hemodialysis? Chest. 2009 Oct;136(4):1128-1133. doi: 10.1378/chest.09-0730. PMID 19809054
- [Background] Shah M, Avgil Tsadok M, Jackevicius CA, Essebag V, Eisenberg MJ, Rahme E, Humphries KH, Tu JV, Behlouli H, Guo H, Pilote L. Warfarin use and the risk for stroke and bleeding in patients with atrial fibrillation undergoing dialysis. Circulation. 2014 Mar 18;129(11):1196-203. doi: 10.1161/CIRCULATIONAHA.113.004777. Epub 2014 Jan 22. PMID 24452752
- [Background] Marinigh R, Lane DA, Lip GY. Severe renal impairment and stroke prevention in atrial fibrillation: implications for thromboprophylaxis and bleeding risk. J Am Coll Cardiol. 2011 Mar 22;57(12):1339-48. doi: 10.1016/j.jacc.2010.12.013. PMID 21414530
- [Background] Skanes AC, Healey JS, Cairns JA, Dorian P, Gillis AM, McMurtry MS, Mitchell LB, Verma A, Nattel S; Canadian Cardiovascular Society Atrial Fibrillation Guidelines Committee. Focused 2012 update of the Canadian Cardiovascular Society atrial fibrillation guidelines: recommendations for stroke prevention and rate/rhythm control. Can J Cardiol. 2012 Mar-Apr;28(2):125-36. doi: 10.1016/j.cjca.2012.01.021. PMID 22433576
- [Background] January CT, Wann LS, Alpert JS, Calkins H, Cigarroa JE, Cleveland JC Jr, Conti JB, Ellinor PT, Ezekowitz MD, Field ME, Murray KT, Sacco RL, Stevenson WG, Tchou PJ, Tracy CM, Yancy CW; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2014 AHA/ACC/HRS guideline for the management of patients with atrial fibrillation: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and the Heart Rhythm Society. J Am Coll Cardiol. 2014 Dec 2;64(21):e1-76. doi: 10.1016/j.jacc.2014.03.022. Epub 2014 Mar 28. No abstract available. PMID 24685669
- [Background] Sood MM, Larkina M, Thumma JR, Tentori F, Gillespie BW, Fukuhara S, Mendelssohn DC, Chan K, de Sequera P, Komenda P, Rigatto C, Robinson BM. Major bleeding events and risk stratification of antithrombotic agents in hemodialysis: results from the DOPPS. Kidney Int. 2013 Sep;84(3):600-8. doi: 10.1038/ki.2013.170. Epub 2013 May 15. PMID 23677245
- [Background] Clase CM, Holden RM, Sood MM, Rigatto C, Moist LM, Thomson BK, Mann JF, Zimmerman DL. Should patients with advanced chronic kidney disease and atrial fibrillation receive chronic anticoagulation? Nephrol Dial Transplant. 2012 Oct;27(10):3719-24. doi: 10.1093/ndt/gfs346. PMID 23114898
- [Background] Gebuis EP, Rosendaal FR, van Meegen E, van der Meer FJ. Vitamin K1 supplementation to improve the stability of anticoagulation therapy with vitamin K antagonists: a dose-finding study. Haematologica. 2011 Apr;96(4):583-9. doi: 10.3324/haematol.2010.035162. Epub 2010 Dec 29. PMID 21193422
- [Background] Sconce E, Avery P, Wynne H, Kamali F. Vitamin K supplementation can improve stability of anticoagulation for patients with unexplained variability in response to warfarin. Blood. 2007 Mar 15;109(6):2419-23. doi: 10.1182/blood-2006-09-049262. Epub 2006 Nov 16. PMID 17110451
- [Background] Cushman M, Booth SL, Possidente CJ, Davidson KW, Sadowski JA, Bovill EG. The association of vitamin K status with warfarin sensitivity at the onset of treatment. Br J Haematol. 2001 Mar;112(3):572-7. doi: 10.1046/j.1365-2141.2001.02635.x. PMID 11260056
- [Background] Sconce E, Khan T, Mason J, Noble F, Wynne H, Kamali F. Patients with unstable control have a poorer dietary intake of vitamin K compared to patients with stable control of anticoagulation. Thromb Haemost. 2005 May;93(5):872-5. doi: 10.1160/TH04-12-0773. PMID 15886802
- [Background] Holbrook A, Schulman S, Witt DM, Vandvik PO, Fish J, Kovacs MJ, Svensson PJ, Veenstra DL, Crowther M, Guyatt GH. Evidence-based management of anticoagulant therapy: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest. 2012 Feb;141(2 Suppl):e152S-e184S. doi: 10.1378/chest.11-2295. PMID 22315259
- [Background] Lam J, Schulman S, Witt DM, Vandvik PO, Qayyum F, Holbrook AM. Anticoagulation control with daily low-dose vitamin k to reduce clinically adverse outcomes and international normalized ratio variability: a systematic review and meta-analysis. Pharmacotherapy. 2013 Nov;33(11):1184-90. doi: 10.1002/phar.1302. Epub 2013 Jun 6. PMID 23744743
- [Background] Rombouts EK, Rosendaal FR, Van Der Meer FJ. Daily vitamin K supplementation improves anticoagulant stability. J Thromb Haemost. 2007 Oct;5(10):2043-8. doi: 10.1111/j.1538-7836.2007.02715.x. Epub 2007 Jul 31. PMID 17666020
- [Background] Westenfeld R, Krueger T, Schlieper G, Cranenburg EC, Magdeleyns EJ, Heidenreich S, Holzmann S, Vermeer C, Jahnen-Dechent W, Ketteler M, Floege J, Schurgers LJ. Effect of vitamin K2 supplementation on functional vitamin K deficiency in hemodialysis patients: a randomized trial. Am J Kidney Dis. 2012 Feb;59(2):186-95. doi: 10.1053/j.ajkd.2011.10.041. Epub 2011 Dec 9. PMID 22169620
- [Background] Cranenburg EC, Schurgers LJ, Uiterwijk HH, Beulens JW, Dalmeijer GW, Westerhuis R, Magdeleyns EJ, Herfs M, Vermeer C, Laverman GD. Vitamin K intake and status are low in hemodialysis patients. Kidney Int. 2012 Sep;82(5):605-10. doi: 10.1038/ki.2012.191. Epub 2012 May 30. PMID 22648294
- [Background] Krueger T, Schlieper G, Schurgers L, Cornelis T, Cozzolino M, Jacobi J, Jadoul M, Ketteler M, Rump LC, Stenvinkel P, Westenfeld R, Wiecek A, Reinartz S, Hilgers RD, Floege J. Vitamin K1 to slow vascular calcification in haemodialysis patients (VitaVasK trial): a rationale and study protocol. Nephrol Dial Transplant. 2014 Sep;29(9):1633-8. doi: 10.1093/ndt/gft459. Epub 2013 Nov 26. PMID 24285427
- [Background] Ford SK, Misita CP, Shilliday BB, Malone RM, Moore CG, Moll S. Prospective study of supplemental vitamin K therapy in patients on oral anticoagulants with unstable international normalized ratios. J Thromb Thrombolysis. 2007 Aug;24(1):23-7. doi: 10.1007/s11239-007-0014-z. Epub 2007 Feb 24. PMID 17323135
- [Background] Reese AM, Farnett LE, Lyons RM, Patel B, Morgan L, Bussey HI. Low-dose vitamin K to augment anticoagulation control. Pharmacotherapy. 2005 Dec;25(12):1746-51. doi: 10.1592/phco.2005.25.12.1746. PMID 16305294
- [Background] Majeed H, Rodger M, Forgie M, Carrier M, Taljaard M, Scarvelis D, Gonsalves C, Rodriguez RA, Wells PS. Effect of 200muG/day of vitamin K1 on the variability of anticoagulation control in patients on warfarin: a randomized controlled trial. Thromb Res. 2013 Sep;132(3):329-35. doi: 10.1016/j.thromres.2013.07.019. Epub 2013 Jul 29. PMID 23953594
- [Background] Schurgers LJ, Shearer MJ, Hamulyak K, Stocklin E, Vermeer C. Effect of vitamin K intake on the stability of oral anticoagulant treatment: dose-response relationships in healthy subjects. Blood. 2004 Nov 1;104(9):2682-9. doi: 10.1182/blood-2004-04-1525. Epub 2004 Jul 1. PMID 15231565
- [Background] Schulman S, Angeras U, Bergqvist D, Eriksson B, Lassen MR, Fisher W; Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medicinal products in surgical patients. J Thromb Haemost. 2010 Jan;8(1):202-4. doi: 10.1111/j.1538-7836.2009.03678.x. Epub 2009 Oct 30. PMID 19878532
- [Background] White HD, Gruber M, Feyzi J, Kaatz S, Tse HF, Husted S, Albers GW. Comparison of outcomes among patients randomized to warfarin therapy according to anticoagulant control: results from SPORTIF III and V. Arch Intern Med. 2007 Feb 12;167(3):239-45. doi: 10.1001/archinte.167.3.239. PMID 17296878
- [Background] Juurlink DN. Drug interactions with warfarin: what clinicians need to know. CMAJ. 2007 Aug 14;177(4):369-71. doi: 10.1503/cmaj.070946. No abstract available. PMID 17698826